CLINICAL TRIAL: NCT01291693
Title: Testing Delivery Channels of Brief Motivational Alcohol Intervention Among General Hospital Inpatients With Risky Drinking: Personal Counseling Versus Computer-generated Feedback Letters
Brief Title: Testing Delivery Channels of Brief Motivational Alcohol Intervention
Acronym: PECO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Principal Investigator, Dr. Jennis Freyer-Adam, Principle investigator, University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108376; DM8-IESO03 (Registry Identifier: University Medicine Greifswald); 108376 (Other Grant/Funding Number: German Cancer Aid); DM8-IESO04 (Registry Identifier: University Medicine Greifswald); 109737 (Other Grant/Funding Number: German Cancer Aid); 110676 (Other Grant/Funding Number: German Cancer Aid); 110543 (Other Grant/Funding Number: German Cancer Aid); 111346 (Other Grant/Funding Number: German Cancer Aid)
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hazardous Drinking
Keywords: Hazardous drinking; general hospital; brief intervention; Motivational Interviewing; computer-generated feedback; stage-tailored; delivery channel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Personal counseling (Experimental)
  Interventions: Behavioral: Personal Counseling
- Computer generated feedback letters (Experimental)
  Interventions: Behavioral: Computer-generated feedback letters
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Personal Counseling — At three time-points, participants receive counseling by health professionals trained in Motivational Interviewing based counseling. To assure that both interventions do not differ in their content, individual manuals generated by a software program are used. Counseling will be face-to-face during the hospital stay, and by phone one and three months later.
  Arms: Personal counseling
Behavioral: Computer-generated feedback letters — At three time points, participants receive feedback letters, tailored to the stages of change according to the TTM, and generated by a computer software program. The first letter is handed out during their hospital stay and includes normative feedback. One and three months later, participants receive ipsative feedback letters by mail.
  Arms: Computer generated feedback letters

SUMMARY:
The aim of this study is to investigate whether motivation-tailored alcohol interventions are more effective when delivered by person or by computer-generated feedback letters. A sample of 920 general hospital inpatients with risky drinking will be recruited through a computerized screening procedure. Patients with more severe alcohol problems will be excluded from the study. Participants will be allocated by time frame randomization to one of three study arms: (1) personal counseling based on Motivational Interviewing, (2) computer-expert system intervention that generates individualized feedback-letters, and (3) control group (treatment-as-usual). The interventions differ in their channel of delivery, but not regarding their content. Both intervention groups receive interventions at three time points: directly after the baseline-assessment at the general hospital, and 1 and 3 months later by mail and phone, respectively. Outcome will be assessed six, 12, 18 and 24 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* General hospital inpatients with risky drinking (AUDIT-C >= 4/5 (women/men) and AUDIT < 20)

Exclusion Criteria:

* Patients already recruited during an earlier hospital stay
* Patients physically and mentally not capable of participating in the study
* Patients with a hospital stay of less than 24 hours
* Patients with insufficient language/ reading skills
* Patients employed at one of the departments participating in the study or conducting the study
* Patients with more severe alcohol problems (AUDIT >= 20)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 975 (Actual)
Dates: Start 2011-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Risky drinking | 6, 12, 18, 24 months
  Determined by using average alcohol consumption per day, heavy occasional drinking, highest blood alcohol concentration, the Alcohol Use Disorder Identification Test-Consumption (AUDIT-C) score

SECONDARY OUTCOMES:
Motivation to reduce drinking | 6, 12, 18, 24 months
  Assessed by a stages of change-algorithm
Attempts to reduce drinking | 6, 12, 18, 24 months
Knowledge about drinking limits | 6, 12, 18, 24 months
Self-efficacy scores | 6 months
  Assessed by a modified short-form of the Alcohol-Abstinence-Self-Efficacy-Scale (AASE). The modified form assesses self-efficacy regarding compliance with drinking limits.
Decisional balance scores | 6 months
  Assessed by a short form of the Alcohol Decisional Balance Scale (ADBS)
Self-rated health | 6, 12, 18, 24 months
Health care utilization | 6, 12, 18, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennis Freyer-Adam, PhD, Principal Investigator — Institute of Social Medicine and Prevention, University Medicine Greifswald; Beate Gaertner, PhD, Principal Investigator — Department of Epidemiology and Health Monitoring, Robert Koch-Institute Berlin; Ulrich John, Prof PhD, Principal Investigator — Institute of Social Medicine and Prevention, University Medicine Greifswald
Locations (1):
- Institute of Social Medicine and Prevention, University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Krolo-Wicovsky F, Baumann S, Tiede A, Bischof G, John U, Gaertner B, Freyer-Adam J. Do in-person and computer-based brief alcohol interventions reduce tobacco smoking among general hospital patients? Secondary outcomes from a randomized controlled trial. Addict Sci Clin Pract. 2023 Nov 13;18(1):68. doi: 10.1186/s13722-023-00425-7. PMID 37957757
- [Derived] Freyer-Adam J, Baumann S, Bischof G, Staudt A, Goeze C, Gaertner B, John U. Social Equity in the Efficacy of Computer-Based and In-Person Brief Alcohol Interventions Among General Hospital Patients With At-Risk Alcohol Use: A Randomized Controlled Trial. JMIR Ment Health. 2022 Jan 28;9(1):e31712. doi: 10.2196/31712. PMID 35089156
- [Derived] Freyer-Adam J, Noetzel F, Baumann S, Aghdassi AA, Siewert-Markus U, Gaertner B, John U. Behavioral health risk factor profiles in general hospital patients: identifying the need for screening and brief intervention. BMC Public Health. 2019 Nov 29;19(1):1594. doi: 10.1186/s12889-019-7931-6. PMID 31783832
- [Derived] Freyer-Adam J, Baumann S, Haberecht K, Tobschall S, Bischof G, John U, Gaertner B. In-person alcohol counseling versus computer-generated feedback: Results from a randomized controlled trial. Health Psychol. 2018 Jan;37(1):70-80. doi: 10.1037/hea0000556. Epub 2017 Oct 2. PMID 28967769
- [Derived] Baumann S, Gaertner B, Haberecht K, Meyer C, Rumpf HJ, John U, Freyer-Adam J. Does impaired mental health interfere with the outcome of brief alcohol intervention at general hospitals? J Consult Clin Psychol. 2017 Jun;85(6):562-573. doi: 10.1037/ccp0000201. Epub 2017 Mar 23. PMID 28333511